CLINICAL TRIAL: NCT03155074
Title: High-Intensity Training Following Lung Transplantation: a Randomized Controlled Trial
Brief Title: High-Intensity Training Following Lung Transplantation
Acronym: HILT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian School of Sport Sciences (Other)
Responsible Party: Principal Investigator, Michael Durheim, Consultant, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017/399
Record Dates: First submitted 2017-05-10; First posted 2017-05-16 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Lung Transplant; Exercise Training
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Intensity Training (Experimental)
  Interventions: Behavioral: High-intensity training
- Usual Care (No Intervention)

INTERVENTIONS:
Behavioral: High-intensity training — The exercise program will include a cardiovascular warm-up, high intensity interval training and progressive resistance training (PRT). The intervention will focus on high-intensity training, mainly by uphill walking on a treadmill at 80-95 % of the maximal heart rate and PRT in three series at 6-12 RM by leg press, chest press, back extension, seat row, and front raises. During the first four weeks, the patients will be introduced to the program while focusing on safety, techniques and familiarization. The endurance intensity and strength load will then continuously increase based on the patients' improvement, tolerance of dyspnea, and feelings of well-being or fatigue on each exercise day.
  Arms: High-Intensity Training

SUMMARY:
The HILT study is a prospective, single-blinded, randomized controlled trial comparing a high-intensity exercise training intervention with usual care among adult lung transplant recipients. Patients randomized to the training intervention arm will undergo individually tailored high-intensity exercise training (80-95% of maximum heart rate) three hours per week for 20 weeks. Training will be conducted at local fitness centers on a one-on-one basis.

ELIGIBILITY:
Inclusion Criteria:

* Stable medical condition in the opinion of the enrolling investigator
* Able and willing to give informed consent

Exclusion Criteria:

* Expected survival less than 12 months
* Unable to complete a maximal exercise test on a treadmill until exhaustion
* Language barrier that interferes with data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-08-22 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Change in peak oxygen uptake | 0-20 weeks
  Measured by cardiopulmonary exercise test

SECONDARY OUTCOMES:
Change in total body composition (fat, muscle and bone mass) | 0-20 weeks
  Measured by dual-energy x-ray absorptiometry (DEXA)
Change in forced expiratory volume in one second (FEV1) | 0-20 weeks
  Measured by spirometry
Change submaximal exercise capacity | 0-20 weeks
  Measured by 6-minute walk distance
Change in leg strength | 0-20 weeks
  Measured by maximum leg press
Change in upper body strength | 0-20 weeks
  Measured by maximum breast press
Change in hand strength | 0-20 weeks
  Measured by grip strength dynamometer
Change in health-related quality of life | 0-20 weeks
  Measured by Short Form 36 (SF-36)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Edvardsen, PhD, Principal Investigator — Oslo University Hospital, Norwegian School of Sport Sciences; Michael T Durheim, MD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gutierrez-Arias R, Martinez-Zapata MJ, Gaete-Mahn MC, Osorio D, Bustos L, Melo Tanner J, Hidalgo R, Seron P. Exercise training for adult lung transplant recipients. Cochrane Database Syst Rev. 2021 Jul 20;7(7):CD012307. doi: 10.1002/14651858.CD012307.pub2. PMID 34282853